CLINICAL TRIAL: NCT03449875
Title: A Post-Market Surveillance Clinical Registry of the TREOVANCE® Stent-Graft for Patients With Infrarenal Abdominal Aortic Aneurysms
Brief Title: Global Post-market Registry for the Treovance Stent-graft.
Acronym: RATIONALE
Status: Completed | Type: Observational
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IP-0024-17
Record Dates: First submitted 2018-01-09; First posted 2018-02-28 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TREOVANCE® Stent-Graft with Navitel® Delivery System — Endovascular repair of abdominal aortic aneurysms.

SUMMARY:
Patients with abdominal aortic aneurysms (AAA) suitable for endovascular aortic repair (EVAR) with Treovance were eligible to participate. Main inclusion criteria were: age 18-85 years; infrarenal AAA without significant infrarenal or distal iliac landing neck calcification or thrombus formation; infrarenal or distal iliac landing neck size requirements specified in the instructions for use. Main exclusion criteria: dissection/ruptured aneurysm or prior AAA endovascular or surgical repair. The primary endpoints were standard EVAR criteria.

DETAILED DESCRIPTION:
The goal of the registry was to collect clinical data of TREOVANCE® device in subjects with infrarenal aortic aneurysms, specifically to evaluate if the diseased pathology is treated with an acceptable technical success rate, an acceptable complication rate and that the device performs as expected.

The following endovascular measures/parameters were assessed for preliminary performance at the follow-up intervals: delivery/deployment, stent-graft migration, stent-graft patency, stent-graft integrity, endoleak, aneurysm sac size changes, limb ischemia, and vascular access complications.

This registry was a prospective, multi-center, post-market non-randomized study. The goal was to gather safety and performance data on the device. Subjects diagnosed with infrarenal aortic aneurysms enrolled into the registry were treated with the TREOVANCE® Stent-Graft with Navitel® Delivery System. Pre-procedure baseline data was gathered as well as post-procedure assessments prior to hospital discharge and 1, 6, and 12 months post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between the ages of 18 and 85.
* Subject must be diagnosed with an infrarenal abdominal aortic aneurysm (AAA), with or without iliac artery involvement, by CT with contrast performed within 3 months of planned implant procedure.
* Subject must have an infrarenal AAA that i. is > 4.5 cm in diameter for females and > 5 cm for males. ii. has increased in diameter by 0.5 cm in the last 6 months
* Subject must have i. infrarenal landing neck length of 10 mm or greater and an angle of less than 60 degrees relative to the long axis of the aneurysm (centerline at lowest renal to centerline at bifurcation) and a suprarenal neck angle of less than 45 degrees relative to the infrarenal neck axis and an inside diameter of 17 mm - 32 mm, or ii. infrarenal landing neck length of 15 mm or greater and an angle of between 60 and 75 degrees relative to the long axis of the aneurysm and a suprarenal neck angle of less than 45 degrees relative to the infrarenal neck axis and an inside diameter of 16 mm-30 mm
* Subject's infrarenal landing neck must i. have no significant calcification or thrombus formation, and ii. meet the vessel size requirements specified in the instructions for use (IFU) for the corresponding devices
* Subject must have lowest renal artery at least 9 cm from the aortic bifurcation
* Subject must have a distal iliac landing neck with i. an inside diameter of 7 mm - 13 mm and a length of at least 10 mm, or ii. an inside diameter of >13 mm - 20 mm and a length of at least 15 mm
* Subject's distal iliac landing neck must i. have no significant calcification or thrombus formation, and ii. meet the vessel size requirements specified for the corresponding devices in the IFU
* Subject must have a total treatment length of at least 13 cm
* Subject must be willing and able to comply with 1-month, 6-month, and 12-month follow-up visits.
* Subject must have adequate vascular access (e.g., patent iliac or femoral arteries) for introduction of the Navitel® Delivery System which is 18F (6 mm) or 19F (6.3 mm) outer diameter based on size of device used. Alternatively, subject's anatomy is suitable for creation of an iliac conduit.
* Subject or Legally Authorized Representative (LAR) must agree to sign hospital issued Informed Consent Form

Exclusion Criteria:

* Subject is pregnant or lactating
* Subject has a dissection or a ruptured aneurysm (as determined by treating physician).
* Subject has a patent inferior mesenteric artery that cannot be sacrificed and an occluded or stenotic celiac and/or superior mesenteric artery
* Implant procedure as planned does not allow for at least one patent hypogastric artery left intact, unless both are occluded on pre-op imaging
* Subject has a lesion that cannot be crossed by a guide wire
* Proximal neck cannot increase by more than 20% over 15 mm; i.e., no conical necks
* Subject has severe untreated coronary artery disease and/or unstable angina, significant areas of myocardium at risk (based on coronary angiogram or radionuclide scans), left ventricular ejection fraction < 20%, or recent diagnosis of CHF
* Subject has had a stroke or MI within 6 months of the planned treatment date
* Subject has chronic obstructive pulmonary disease requiring routine need for oxygen therapy outside the hospital setting (e.g., daily or nightly home use)
* Subject has an active systemic infection or is suspected of having an active systemic infection (e.g., AIDS/HIV, sepsis)
* Subject is morbidly obese (more than 100% over the ideal body weight or as defined by institutional standards) or has other clinical conditions that severely compromise or impair x-ray visualization of the aorta
* Subject has significant or circumferential mural thrombus in the proximal aortic neck
* Subject has a blood coagulation disorder or bleeding diathesis the treatment for which cannot be suspended pre- and post-repair
* Subject is in acute or chronic renal failure (creatinine > 2.5 mg/dL)
* Subject has less than two-year life expectancy as evidenced by factors prohibiting major medical intervention (e.g., presence of malignancy, severe cardiopulmonary disease, etc.)
* Subject is participating in another research study, has received investigational study drug within 30 days of planned procedure, or has received an investigational device within one year of planned procedure.
* Subject is confronted with other medical, social or psychological issues that the investigator believes may interfere with study treatment or follow-up. These reasons must be documented. An example may include adherence to a theological or personal doctrine with aversion or opposition to blood transfusion.
* Subject has had a prior AAA repair (endovascular or surgical)
* Subject has an untreatable allergy or sensitivity to contrast media, nitinol/nickel, or polyester
* Subject has undergone other major surgical or medical intervention within 45 days of the planned procedure or is planning to undergo other major surgical or medical intervention within 45 days post implantation (e.g., CABG, organ transplantation, renal stenting, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with infrarenal aortic aneurysms requiring endovascular repair.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting Major Adverse Events | Through 12 months
  Primary safety outcome will be assessed by measurement of mortality and major morbidity rates through reporting of the following events:
  * Death
  * Stroke
  * Myocardial Infarction
  * Renal Failure requiring renal replacement therapy
  * Respiratory Failure, defined as ventilator-dependent
  * Paraparesis / Paraplegia (excludes paraparesis)
  * Bowel ischemia
  * Treated aneurysm rupture

SECONDARY OUTCOMES:
Rate of Device Delivery/Deployment Success | Procedure / Study Day 0
  Device effectiveness will be measured through the rate of successful delivery and deployment during the index procedure
Rate of Stent-Graft Migration greater than 10mm | 6 months and 12 months
  Device effectiveness will be measured by the rate of Stent-Graft Migration greater than 10mm as compared to the first post procedure imaging
Rate of Stent-Graft Patency | 1 month, 6 months and 12 months
  Device effectiveness will be measured by the rate of Stent-Graft Patency observed
Rate of Stent-Graft Integrity | 1 month, 6 months and 12 months
  Device effectiveness will be measured by the rate of Stent-Graft Integrity observed
Rate of Endoleaks | 1 month, 6 months and 12 months
  Device effectiveness will be measured by the rate of Endoleaks reported
Rate of Aneurysm Sac Size Changes | 6 months and 12 months
  Device effectiveness will be measured by the rate of Aneurysm Sac Size Changes at 6 months and 12 months as compared to the first post-procedure imaging
Rate of Limb Ischemia | 1 month, 6 months and 12 months
  Device effectiveness will be measured by the rate of Limb Ischemia resulting in limb loss
Rate of Vascular Access Complications | 1 month, 6 months and 12 months
  Device effectiveness will be measured by the rate of Vascular Access Complications
Rate of unintentional covering of renal arteries and / or hypogastric arteries | Procedure / Study Day 0
  Device effectiveness will be measured by the rate of unintentional covering of renal arteries and / or hypogastric arteries during the index procedure

OTHER OUTCOMES:
Summary results of procedural data and outcomes | 1 month, 6 months and 12 months
  Procedural data and outcomes will be summarized descriptively, including:
  * Type of anesthesia
  * Duration of procedure time (first cut to last stitch)
  * Time in ICU
  * Duration of hospitalization
  * Volume of blood loss
  * Volume of blood replaced
  * Subjects requiring blood transfusion
  * Type of arterial access (percutaneous, cut down)
  * Reinterventions

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Setacci, MD, PhD, Study Chair — Department of Medicine, Surgery and Neuroscience, University of Siena Viale Bracci 1, 53100 Siena, Italy
Locations (32):
- Chile (2):
  - Hospital Barros Luco Trudeau, Santiago
  - Hospital de la Dirección de Previsión de Carabineros de Chile, Santiago
- Rigshospitalet, National Hospital and University of Copenhagen, Copenhagen, Denmark
- Germany (4):
  - Deutsches Herzzentrum Berlin, Berlin
  - Bonifatius Hospital, Lingen
  - Theresienkrankenhaus und St. Hedwig-Klinik, Mannheim
  - Universitätsklinikum Tübingen, Tübingen
- Greece (2):
  - Evaggelismos General Hospital, Athens
  - Georgios Gennimatas Thessaloniki General Hospital, Thessaloniki
- Queen Mary Hospital, University of Hong Kong, Hong Kong, Hong Kong
- Semmelweis Medical University Budapest, Budapest, Hungary
- Cork University Hospital, Cork, Ireland
- Italy (3):
  - Casa Di Cura Villa Dei Fiori, Acerra
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
- Netherlands (2):
  - ZiekenhuisGroep Twente, Almelo
  - Universitair Medisch Centrum Utrecht, Utrecht
- Haukeland University Hospital, Bergen, Norway
- Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin, Poland
- Spain (5):
  - Hospital HM Modelo, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Solna
- Lampang Hospital, Lampang, Thailand
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge University Hospitals, Cambridge
  - Manchester Royal Infirmary, Central Manchester University Hospitals, Manchester
  - John Radcliffe Hospital, Oxford University Hospitals, Oxford
- Instituto Urológico San Román, Caracas, Venezuela
- Cho Ray Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Murray D, Szeberin Z, Benevento D, Abdallah F, Palasciano G, Lescan M, Uberoi R, Setacci C. A comparison of clinical outcomes of abdominal aortic aneurysm patients with favorable and hostile neck angulation treated by endovascular repair with the Treovance stent graft. J Vasc Surg. 2020 Jun;71(6):1881-1889. doi: 10.1016/j.jvs.2019.07.096. Epub 2019 Nov 2. PMID 31690524
- [Derived] Uberoi R, Setacci C, Lescan M, Lorido A, Murray D, Szeberin Z, Zubilewicz T, Riambau V, Chartrungsan A, Tessarek J; RATIONALE Investigators. Global Post-Market Clinical Follow-up of the Treovance Stent-Graft for Endovascular Aneurysm Repair: One-Year Results From the RATIONALE Registry. J Endovasc Ther. 2018 Dec;25(6):726-734. doi: 10.1177/1526602818803939. Epub 2018 Oct 3. PMID 30280649